CLINICAL TRIAL: NCT03870152
Title: Electrocautery Ablation for the Prevention of Lung Cancer
Acronym: EARL
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: This decision was made due to lower than expected recruitment levels into the trial
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UCL/12/1585
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Lung Cancer Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EC treatment (Intervention Arm) (Experimental): Patients in the intervention arm will receive up to three rounds of EC treatment (no more than one round annually) to all their HGLs identified at baseline. Follow-up is the same as for Control Arm patients: a bronchoscopy surveillance visit at 6, 12, 24, and at 36 months post-randomisation; with further bronchoscopy surveillance visits at 18 and/or at 30 months post-randomisation (dependent on lesion appearance).
  Interventions: Procedure: Electrocautery Ablation (EC)
- AFB Surveillance (Control Arm) (No Intervention): Patients randomised to the surveillance (Control Arm) will have: bronchoscopy surveillance at 6, 12, 24, and at 36 months post-randomisation; with further bronchoscopy surveillance visits at 18 and/or at 30 months post-randomisation (dependent on lesion appearance).

INTERVENTIONS:
Procedure: Electrocautery Ablation (EC) — For the purposes of the trial, one round of EC treatment consists of two individual EC treatments with a post-EC bronchoscopy in between to check for a response to the 1st EC treatment. Within each round, the second EC treatment will only be administered if the post-treatment bronchoscopy confirms presence of persistent high grade disease. Patients in the intervention arm will receive up to three rounds of EC treatment (no more than one round annually) to all their HGLs identified at baseline.
  Arms: EC treatment (Intervention Arm)

SUMMARY:
This study evaluates whether EC treatment is effective in delaying the progression of high-grade lung lesion(s) to invasive lung cancer. Participants will be randomised to receive either electrocautery (EC) treatment with bronchoscopy surveillance (=intervention), or bronchoscopy surveillance alone (=control) in a 2:1 ratio.

DETAILED DESCRIPTION:
Squamous cell carcinoma of the lung develops through a transition of progressive cytological aberration, from normal to metaplasia, mild, moderate, and severe dysplasia and then carcinoma in situ (CIS) before becoming an invasive cancer. Progression rates to invasive carcinoma can vary depending on the initial grade of the lesion and it is generally accepted that high-grade lesions are more likely to progress to invasive cancer than low-grade lesions. Early detection and treatment of these lesions is critical to improving survival. There is no evidence base examining how, or whether these high-grade lesions (HGLs) should be treated, resulting in diverse treatment practices both nationally and internationally. This is the first randomised clinical trial of a bronchoscopic intervention in treating HGLs using EC.

EARL is a phase II/III multicentre 2:1 randomised controlled trial to evaluate the effectiveness of electrocautery (EC) in the treatment of high-grade lesions of the lung. All patients consented/registered onto the trial will have an bronchoscopy (AFB or NBI) to check for high-grade lesions (HGLs) in the lung, as verified by tissue biopsy. Only patients with ≥1 lung histologically confirmed lung HGL will be randomised to receive either electrocautery ablation (EC) treatment and bronchoscopy surveillance (= intervention), or bronchoscopy surveillance (= control).

The principal objective of the main phase II trial is to demonstrate that airway High-Grade Lesions (HGLs) that are treated with electrocautery are less likely to progress to lung cancer compared to HGLs that are not treated with electrocautery.

ELIGIBILITY:
Inclusion criteria:

1. Patients with ≥1 airway HGL (defined as severe dysplasia or carcinoma in situ on histology)

   PRE-REGISTRATION

   Patient has a high likelihood of having airway HGLs as evaluated by investigator:
   * patient already part of existing surveillance programme or
   * HGL identified at other hospital and patient is referred to study site or
   * patient has abnormal sputa and patient is referred to study site

   PRE-RANDOMISATION Following registration, patients undergo a baseline bronchoscopy and only those with ≥1 airway HGL(s) can continue to randomisation provided they continue to meet all the inclusion/exclusion criteria below
2. Absence of primary lung cancer as confirmed by CT thorax OR recent surgical removal of a lung cancer with clear resection margins (of cancer) confirmed OR recent successful curative SABR treatment, as confirmed by MDT
3. Male or female patients ≥18 years of age
4. No upper age limit but life expectancy thought to be at least 3 years (in the opinion of the treating clinician)
5. ECOG Performance Score 0-2
6. FEV1 ≥ 25% of predicted*
7. DLCO/TLCO ≥ 20% of predicted (only required for registration)*
8. Patients who are women of child-bearing potential (WOCBP) must also have a negative pregnancy test at the following time points:

   * One pregnancy test prior to registration
   * One pregnancy test within 24 hours prior to the 1st EC treatment within each EC treatment round
9. Consent to donation of biological samples for translational work. Patients will be deemed ineligible if they do not consent to donate translational samples
10. Patient is willing and able to comply to protocol procedures and attend all study visits including all bronchoscopy and EC treatment visits.

    * if spirometry is not possible (e.g. due to COVID-19) investigator assessment that the patient is sufficiently fit for bronchoscopy and EC treatment is permissible.

Exclusion criteria:

1. Finding of (micro)-invasive disease on histology (assessed at randomisation)
2. Patients who have one or more HGL present for ≥5 years which have remained persistent on white light or autofluorescence bronchoscopy (AFB) surveillance
3. Detection of active cancer or on systemic treatment for cancer, excluding basal cell skin cancers
4. Previous radiotherapy to the treatment area
5. ECOG Performance Score >2
6. Patients who have one or more HGL greater than 3cm in length
7. Patients with a history of pulmonary hypertension
8. Patients who are anticoagulated for prosthetic heart valves
9. Decompensated heart disease with life expectancy less than 3 years
10. Severe liver and renal insufficiency with life expectancy less than 3 years
11. Patient unlikely to cooperate with a 3-year follow-up; medical or psychological condition at the discretion of the investigator which would not permit compliance with the protocol or meaningful signed informed consent
12. Participation in another study with an investigational medicinal product within one month prior to registration
13. Pregnant patients (confirmed by serum/urine ß-HCG)
14. Any other known condition which is assessed as an intolerable risk by the investigator upon inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
The time to progression of any index HGL in a patient within a 3-year follow up (phase II and III) | 3 years post randomisation
  The time to progression of any index HGL in a patient to invasive lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: EARL Trial Coordinator, Study Chair — UCL
Locations (1):
- UCLH, London, United Kingdom